CLINICAL TRIAL: NCT06629532
Title: The REgistry Study on Multimodality trEAtment foR Cerebral Hemorrhage
Acronym: RESEARCH
Status: Not yet recruiting | Type: Observational
Sponsor: Tao Liu (Other)
Collaborators: Tianjin Medical University General Hospital (Other); Xuanwu Hospital, Beijing (Other)
Responsible Party: Sponsor-Investigator, Tao Liu, MD, The George Institute
Organization: The George Institute (Other)
Other Study IDs: Thegeorgeinstitute; 82071390 (Other Grant/Funding Number: National Natural Science Foundation of China); 82271394 (Other Grant/Funding Number: National Natural Science Foundation of China); 8247050928 (Other Grant/Funding Number: National Natural Science Foundation of China)
Record Dates: First submitted 2024-10-03; First posted 2024-10-08 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-10

CONDITIONS: Intracerebral Hemorrhage
Keywords: intracerebral hemorrhage; Outcome; Management; Surgical interventions; Real-world; Disparities; Multicentric data
MeSH Terms: conditions — Cerebral Hemorrhage | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: medical management, surgical interventions, and rehabilitative strategies — By leveraging a wide array of treatment data - including medical management, surgical interventions, and rehabilitative strategies - the RESEARCH registry intends to provide a granular view of current treatment landscapes and their direct impact on patient recovery and quality of life.

SUMMARY:
The REgistry Study on multimodality trEAtment foR Cerebral Hemorrhage (RESEARCH) aims to address these challenges by establishing a comprehensive national registry. This initiative will collect detailed, longitudinal data on the clinical characteristics, treatment modalities, and outcomes of patients with ICH across various regions. By leveraging a wide array of treatment data - including medical management, surgical interventions, and rehabilitative strategies - the RESEARCH registry intends to provide a granular view of current treatment landscapes and their direct impact on patient recovery and quality of life.

DETAILED DESCRIPTION:
Cerebral hemorrhage, also known as intracerebral hemorrhage (ICH), is a severe neurological condition characterized by abrupt bleeding within the brain tissues, leading to high rates of mortality and morbidity worldwide. In China, where the burden of cerebrovascular diseases is substantial due to the aging population and prevalence of risk factors such as hypertension and diabetes, the impact of ICH is particularly pronounced. Despite advancements in medical science, the prognosis for patients suffering from ICH remains poor, with a high proportion of survivors experiencing significant disability.

Current treatment protocols for ICH involve a range of strategies, from conservative management to surgical interventions. However, the heterogeneity in clinical practices and patient responses highlights a significant gap in standardized treatment efficacy.

This registry study is not only pivotal for enhancing the understanding of effective treatment combinations but also crucial for identifying potential disparities in the application of treatment modalities across different healthcare settings. Through the analytical power of this large-scale, multicentric data, RESEARCH will contribute significantly to optimizing treatment paradigms and ultimately, shaping policy changes that aim to reduce the mortality and enhance the recovery rates of patients suffering from cerebral hemorrhage.

There is an urgent need to evaluate these multimodal treatment approaches on a broader scale to understand their real-world effectiveness and develop guidelines that can be systematically applied to improve patient outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Cerebral hemorrhage

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Cerebral hemorrhage from various causes
Sampling Method: Non-Probability Sample
Enrollment: 100000 (Estimated)
Dates: Start 2024-10-15 (Estimated); Primary Completion 2044-10-15 (Estimated); Study Completion 2049-10-15 (Estimated)

PRIMARY OUTCOMES:
modified Rankin Score (mRS) | at least 6 months
  0=no symptoms, 1=no significant disability, 2=slight disability, 3= moderate disability, 4=moderate severe disability, 5=severe disability, 6=death

IPD SHARING:
Plan to Share IPD: Undecided